CLINICAL TRIAL: NCT00110266
Title: An Open Label, Safety and Tolerability Study of Deferasirox for Treatment of Transfusional Iron Overload in Low-risk and INT-1, Myelodysplastic Patients Using Serum Ferritin Monitoring
Brief Title: Study of Deferasirox for Treatment of Transfusional Iron Overload in Myelodysplastic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670AUS03; NCT00343837 (obsolete NCT alias)
Record Dates: First submitted 2005-05-04; First posted 2005-05-05 (Estimated); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Myelodysplastic Syndrome; Iron Overload
Keywords: ICL670; Deferasirox; Iron chelation; Chelator; Desferal
MeSH Terms: conditions — Myelodysplastic Syndromes; Iron Overload | interventions — Deferasirox; Chelating Agents; Deferoxamine; Iron Chelating Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICL670 (Experimental): Evaluate the safety and tolerability of deferasirox 20 mg/kg/day over one year in patients with MDS
  Interventions: Drug: Deferasirox

INTERVENTIONS:
Drug: Deferasirox — 20 mg/kg/day over one year in patients with MDS
  Other Names: ICL670A; chelator; desferal; iron chelation

SUMMARY:
The purpose of this trial is to examine the safety and efficacy of deferasirox in patients with Myelodysplastic Syndrome (MDS) and chronic iron overload from blood transfusions.

DETAILED DESCRIPTION:
Study entry requires a diagnosis of low or intermediate (INT-1) risk MDS per International Prognostic Scoring System (IPSS) criteria and serum ferritin ≥ 1000 ng/mL. Patients must have had at least 30 prior red blood cell transfusions. Deferasirox will be administered at an initial dose of 20 mg/kg orally once per day. Patient transfusion history and at least three complete blood count (CBC) values must be available for the 12 weeks prior to study registration for patients with MDS and chronic iron overload from blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with low or intermediate (INT-1) risk MDS
* Patients can be EITHER naïve to iron chelation OR have had prior treatment with deferoxamine (DFO).
* Age greater than or equal to 18 years
* Availability of transfusion records for the 12 weeks prior to registration
* A lifetime minimum of 30 previous packed red blood cell transfusions
* Availability of at least three CBC values (pretransfusion) during the 12 weeks prior to registration
* Serum Ferritin:

For entry into the screening period, serum ferritin ≥ 1000 ng/mL on at least two occasions, at least two weeks apart, during the prior year.

Serum ferritin ≥ 1000 ng/mL at screening via the central lab.

* Life expectancy ≥ 6 months
* Sexually active women must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months)
* Able to provide written informed consent

Exclusion Criteria:

* Serum creatinine above the upper limit of normal
* Alanine aminotransferase (ALT) > 500 U/L during screening
* Clinical or laboratory evidence of active Hepatitis B or C
* Urinary protein/creatinine ratio > 0.5 mg/mg
* History of HIV positive test result (ELISA or Western blot)
* Eastern Cooperative Oncology Group (ECOG) Performance Status > 2
* Patients with uncontrolled systemic hypertension
* Unstable cardiac disease not controlled by standard medical therapy
* Patients with a diagnosis of or history of clinically relevant ocular toxicity related to iron chelation
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent study treatment
* Pregnancy or breast feeding
* Treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days
* Other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of study drug
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2005-07-25 (Actual); Primary Completion 2008-03-28 (Actual); Study Completion 2008-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (45):
- United States (41):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Mayo Clinic, Phoenix, Arizona
  - Bay Area Cancer Research Group, Concord, California
  - City of Hope National Medical Center, Duarte, California
  - Cedars-Sinai Medical Center, UCLA School of Medicine, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCSF, San Francisco, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Emory University School of Medicine/Winship Cancer Institute, Atlanta, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Novartis Investigative Site, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky College of Medicine, Markey Cancer Center, Lexington, Kentucky
  - Cabrini Center for Cancer Care/Christus St. Frances Cabrini Hospital, Alexandria, Louisiana
  - St. Agnes HealthCare, Baltimore, Maryland
  - Rush Cancer Institute Univ. of Massachussets Medical Center, Worcester, Massachusetts
  - Novartis Investigative Site, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Center for Cancer Care & Research (TCCCR), St Louis, Missouri
  - Oncology Hematology West, PC, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - The Cancer Center at Hackensack University, Hackensack, New Jersey
  - NMOHC, Albuquerque, New Mexico
  - Roswell Park Cancer Center, Buffalo, New York
  - Rochester General Hospital/Lipson Cancer and Blood Center, Rochester, New York
  - Cancer Care of WNC, Asheville, North Carolina
  - Wake Forest UniversitComprehensive Cancer Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Thomas Jefferson University; Jefferson Medical College, Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital Cancer Institute, Pittsburgh, Pennsylvania
  - The West Cancer Clinic, Memphis, Tennessee
  - Novartis Investigative site, Nashville, Tennessee
  - Baylor/The Methodist Hospital, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Arlington Fairfax Hematology Oncology PC, Arlington, Virginia
  - Novartis Investigative Site, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec

REFERENCES:
- [Result] List AF, Baer MR, Steensma DP, Raza A, Esposito J, Martinez-Lopez N, Paley C, Feigert J, Besa E. Deferasirox reduces serum ferritin and labile plasma iron in RBC transfusion-dependent patients with myelodysplastic syndrome. J Clin Oncol. 2012 Jun 10;30(17):2134-9. doi: 10.1200/JCO.2010.34.1222. Epub 2012 Apr 30. PMID 22547607
- See also: Results for CICL670AUS03 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2782
- See also: Publication (Embasse # 2012421150) — https://www.ncbi.nlm.nih.gov/pubmed/?term=22547607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 39 centers in the United States and 6 centers in Canada
Pre-assignment Details: A total of 176 participants enrolled in the study, of these 173 participants were treated. Three of the enrolled participants were not treated as 2 withdrew the consent and 1 died even before initiating the treatment.
  Of the 173 treated participants, 95 completed the study and 78 discontinued treatment prematurely.
Groups:
- Deferasirox: Participants received Deferasirox 20 Milligrams per Kilogram per day (mg/kg/day) orally once per day (OD) for one year. The appropriate daily dose was calculated by participants actual body weight. Deferasirox was taken every morning 30 minutes before breakfast, preferably around the same time between 7:00 and 9:00 AM each day. The tablets was dropped into water or apple juice or orange juice and gently stirred for 1 to 3 minutes until completely dispersed.
Period: Overall Study
Arm/Group | Deferasirox
Started | 173
Completed | 95
Not Completed | 78
Not completed — Adverse Event | 27
Not completed — Abnormal laboratory value | 15
Not completed — Withdrawal by Subject | 16
Not completed — Death | 17
Not completed — Unsatisfactory therapeutic effect | 2
Not completed — Participant condition no longer requires study drug | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) population consisted of all participants who received at least 1 dose of Deferasirox.
Groups:
- Deferasirox: Participants received Deferasirox 20 mg/kg/day orally OD for one year. The appropriate daily dose was calculated by participants actual body weight. Deferasirox was taken every morning 30 minutes before breakfast, preferably around the same time between 7:00 and 9:00 AM each day. The tablets was dropped into water or apple juice or orange juice and gently stirred for 1 to 3 minutes until completely dispersed.
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 159
  Black | 4
  Oriental | 4
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the study, whether or not considered related to the participant's participation in the study. Serious Adverse Events include adverse events that result in either of death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Time Frame: up to 53 Weeks
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
Participants | 171

2. Secondary Outcome: Change in Serum Ferritin From Baseline to Weeks 13, 25, 37 and 53
Description: Change in levels of serum ferritin from baseline to 3, 6, 9 and 12 months (Weeks 13, 25, 37 and 53).
Time Frame: From Baseline to Weeks 13, 25, 37 and 53
Population: The Full Analysis Set (FAS) populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: μg/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 172
μg/L
  Baseline | 2771.5 [863 to 9993]
  Week 13: number analyzed (Participants) | 142
  Week 13 | -146.5 [-6679 to 3260]
  Week 25: number analyzed (Participants) | 124
  Week 25 | -167.5 [-5034 to 2265]
  Week 37: number analyzed (Participants) | 110
  Week 37 | -505.0 [-3699 to 4132]
  Week 53: number analyzed (Participants) | 91
  Week 53 | -592.0 [-5752 to 5948]

3. Secondary Outcome: Change in Labile Plasma Iron (LPI)
Description: LPI represents the component of non-transferrin bound iron and is an indicator of iron overload. The blood sample for LPI determinations was collected at Week 1 (prior to first dose) and at Weeks 13, 25, 37 and 49. LPI was calculated as 1 LPI unit = the quantity of reactive oxygen species produced by approximately 1.5 μM Fe
Time Frame: From Baseline to Weeks 13, 25, 37 and 49
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: LPI Unit
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
LPI Unit
  Baseline: number analyzed (Participants) | 163
  Baseline | 0.30 [0.0 to 3.6]
  Week 13: number analyzed (Participants) | 117
  Week 13 | -0.10 [-3.3 to 2.2]
  Week 25: number analyzed (Participants) | 107
  Week 25 | -0.20 [-2.4 to 1.2]
  Week 37: number analyzed (Participants) | 89
  Week 37 | -0.30 [-3.4 to 0.6]
  Week 49: number analyzed (Participants) | 64
  Week 49 | -0.45 [-3.6 to 0.9]

4. Secondary Outcome: Directly Chelatable Iron (DCI)
Description: The blood sample for DCI determinations were collected at Week 1 (prior to first dose) and at Weeks 13, 25, 37 and 49.
Time Frame: From Baseline to Weeks 13, 25, 37 and 49
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: µM
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
µM
  Baseline: number analyzed (Participants) | 163
  Baseline | 0.00 [0.0 to 1.3]
  Week 13: number analyzed (Participants) | 117
  Week 13 | 0.00 [-0.5 to 2.2]
  Week 25: number analyzed (Participants) | 107
  Week 25 | 0.00 [-0.6 to 2.6]
  Week 37: number analyzed (Participants) | 89
  Week 37 | 0.00 [-0.6 to 1.4]
  Week 49: number analyzed (Participants) | 64
  Week 49 | 0.00 [-0.6 to 1.6]

5. Secondary Outcome: Total Iron Levels
Description: Levels of non-transferrin bound iron (NTBI) and serum iron from baseline to 3,6,9 and 12 months (Weeks 13, 25, 37 and 49) were assessed.
Time Frame: From Baseline to Weeks 13, 25, 37, 49 and 53
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: μg/dL
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
μg/dL
  Baseline | 194.0 [48.0 to 409.0]
  Week 13: number analyzed (Participants) | 140
  Week 13 | 230.50 [54.0 to 863.0]
  Week 25: number analyzed (Participants) | 125
  Week 25 | 222.0 [27.0 to 497.0]
  Week 37: number analyzed (Participants) | 111
  Week 37 | 212.0 [53.0 to 480.0]
  Week 49: number analyzed (Participants) | 92
  Week 49 | 218.0 [48.0 to 929.0]
  Week 53: number analyzed (Participants) | 91
  Week 53 | 221.00 [16.0 to 455.0]

6. Secondary Outcome: Serum Transferrin Levels
Description: Serum transferrin from baseline to 3, 6, 9 and 12 months of treatment (Visit Weeks 13, 25, 37 and 49) were assessed.
Time Frame: From Baseline to Weeks 13, 25, 37, 49 and 53
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
mg/dL
  Baseline: number analyzed (Participants) | 171
  Baseline | 156.0 [83.0 to 244.0]
  Week 13: number analyzed (Participants) | 143
  Week 13 | 161.0 [108.0 to 257.0]
  Week 25: number analyzed (Participants) | 123
  Week 25 | 160.0 [107.0 to 266.0]
  Week 37: number analyzed (Participants) | 110
  Week 37 | 158.0 [88.0 to 272.0]
  Week 49: number analyzed (Participants) | 92
  Week 49 | 160.0 [90.0 to 289.0]
  Week 53: number analyzed (Participants) | 90
  Week 53 | 161.00 [99.0 to 253.0]

7. Secondary Outcome: Transferrin Saturation
Description: Levels of transferrin saturation from baseline to 3, 6, 9 and 12 months.
Time Frame: From Baseline to Weeks 13, 25, 37, 49 and 53
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percentage of saturation
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
percentage of saturation
  Baseline: number analyzed (Participants) | 172
  Baseline | 91.00 [20.0 to 94.0]
  Week 13: number analyzed (Participants) | 139
  Week 13 | -11.00 [-73.0 to 57.0]
  Week 25: number analyzed (Participants) | 124
  Week 25 | -11.00 [-66.0 to 58.0]
  Week 37: number analyzed (Participants) | 110
  Week 37 | -12.50 [-68.0 to 57.0]
  Week 49: number analyzed (Participants) | 91
  Week 49 | -12.00 [-72.0 to 65.0]
  Week 53: number analyzed (Participants) | 89
  Week 53 | -18.00 [-69.0 to 64.0]

8. Secondary Outcome: Transfusion Requirements
Description: Number of participants receiving transfusions, the summarized during the study.
Time Frame: up to 1 year
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
Participants
  Screening: number analyzed (Participants) | 171
  Screening | 163
  Week 1 through 13: number analyzed (Participants) | 147
  Week 1 through 13 | 136
  Week 14 through 26: number analyzed (Participants) | 128
  Week 14 through 26 | 119
  Week 27 through 39: number analyzed (Participants) | 113
  Week 27 through 39 | 98
  Week 40 through 52: number analyzed (Participants) | 83
  Week 40 through 52 | 72

9. Secondary Outcome: Frequency of Hematologic Improvement During the Study
Description: Hematologic responses defined by International Working Group response criteria in myelodysplasia. Hematologic Improvement (HI) responses, at least 9 weeks defined as:
  Erythroid response (pretreatment, <11 g/dL): Hgb increase by 1.5 g/dL; Relevant reduction units of Red blood cell (RBC) transfusions by absolute number at least 4 RBC transfusions/8 week compared with pretreatment transfusion number in previous 8 weeks; Only RBC transfusions for Hgb of 9.0 g/dL pretreatment count in RBC transfusion response evaluation; Platelet response (pretreatment,<100x10^9/L): If starting with >20x10^9/L platelets: absolute increase 30x10^9/L, Increase from baseline <20 x10^9/L to >20x10^9/L and by =/> 100%; Neutrophil response (pretreatment, <1.0x10^9/L): =/> 100% increase & absolute increase >0.5x10^9/L; Progression or relapse after HI: At least 1 of the following: =/>50% decrement from max response levels in granulocytes or platelets; Reduction in Hgb by 1.5 g/dL; or Transfusion dependence.
Time Frame: up to 1 year
Population: The analysis was performed on Per protocol population defined as number of participants who did not present any major deviations from protocol and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 91
Participants
  Response (Yes) | 7
  Response (No) | 74
  Missing | 10

10. Secondary Outcome: Trough Plasma Deferasirox Concentration
Description: The Pharmacokinetic (PK) parameters were assessed at Week 13, 25, 37 and 49 using Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) method.
Time Frame: At Week 13, 25, 37 and 49
Population: The full analysis set populations consisted of all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: μmol/L
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
μmol/L
  Week 13: number analyzed (Participants) | 129
  Week 13 | 21.200 [0.00 to 209.0]
  Week 25: number analyzed (Participants) | 114
  Week 25 | 26.700 [0.00 to 331.0]
  Week 37: number analyzed (Participants) | 99
  Week 37 | 25.200 [0.00 to 242.0]
  Week 49: number analyzed (Participants) | 77
  Week 49 | 30.700 [0.00 to 223.0]

11. Secondary Outcome: Treatment Compliance to Deferasirox
Description: Treatment compliance was assessed using records of study medication used, dosages administered, and intervals between visits during the study. Drug accountability was noted by the field monitor during site visits and at the completion of the trial. Participants were asked to return all unused medication at monthly visits.
Time Frame: up to 1 year
Population: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Measure: Number; unit: participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 173
participants
  20 to < 40 % | 2
  40 - < 60 % | 1
  60 - < 80 % | 4
  80 - < 100 % | 89
  100 - < 120 % | 65
  ≥ 120 % | 12

12. Secondary Outcome: The Prevalence of Hereditary Hemochromatosis Gene (HFE) Gene Mutations
Description: HFE (hemochromatosis) gene mutations in the Myelodysplastic Syndrome (MDS) population, the trial included testing for the C282Y, H63D and S65C HFE gene mutations. One blood sample was collected at Baseline (Week 1), or, if that visit was missing, the sample was taken at Week 13 (Month 3). Only one blood sample was to be taken from each participant.
Time Frame: up to Week 13 (Month 3)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox
Number analyzed (Participants) | 94
Participants
  C282Y: Negative | 85
  C282Y: Positive Heterozygous | 9
  H63D: Negative | 70
  H63D: Positive Heterozygous | 24
  S65C: Negative | 92
  S65C: Positive Heterozygous | 2

ADVERSE EVENTS:
Time Frame: All Adverse Event Were Collected From Start of Treatment up to 53 Weeks
Description: Out of 176 participants enrolled in the study, 173 participants received study medication. As, two participants withdrew consent and one died before initiating the treatment, were not considered for this analysis.
  The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Groups:
- Enrolled, Not Treated: Participant died before initiating the treatment.
Arm/Group | Deferasirox | Enrolled, Not Treated
All-Cause Mortality (participants affected / at risk) | 17/173 | 1/3
Serious Adverse Events (participants affected / at risk) | 78/173 | 0/3
Other Adverse Events (participants affected / at risk) | 166/173 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=173) | Enrolled, Not Treated (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Concomitant disease progression (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 0
Induration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 5 | 0
Pyrexia (General disorders) | 7 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 2 | 0
Clostridium bacteraemia (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 12 | 0
Propionibacterium infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 4 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Lymphorrhoea (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deferasirox (N=173) | Enrolled, Not Treated (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 0
Splenomegaly (Blood and lymphatic system disorders) | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 0
Tachycardia (Cardiac disorders) | 4 | 0
Vision blurred (Eye disorders) | 9 | 0
Abdominal distension (Gastrointestinal disorders) | 16 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 0
Constipation (Gastrointestinal disorders) | 30 | 0
Diarrhoea (Gastrointestinal disorders) | 101 | 0
Dyspepsia (Gastrointestinal disorders) | 17 | 0
Flatulence (Gastrointestinal disorders) | 6 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 60 | 0
Stomach discomfort (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 12 | 0
Vomiting (Gastrointestinal disorders) | 21 | 0
Asthenia (General disorders) | 12 | 0
Chest discomfort (General disorders) | 8 | 0
Chest pain (General disorders) | 9 | 0
Chills (General disorders) | 8 | 0
Fatigue (General disorders) | 68 | 0
Gait disturbance (General disorders) | 5 | 0
Oedema (General disorders) | 6 | 0
Oedema peripheral (General disorders) | 35 | 0
Pain (General disorders) | 9 | 0
Pyrexia (General disorders) | 28 | 0
Bronchitis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 4 | 0
Cystitis (Infections and infestations) | 5 | 0
Infection (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 16 | 0
Pneumonia (Infections and infestations) | 9 | 0
Sinusitis (Infections and infestations) | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 19 | 0
Urinary tract infection (Infections and infestations) | 17 | 0
Contusion (Injury, poisoning and procedural complications) | 14 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 5 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Blood creatinine increased (Investigations) | 34 | 0
Blood urea increased (Investigations) | 4 | 0
International normalised ratio increased (Investigations) | 4 | 0
Weight decreased (Investigations) | 12 | 0
Anorexia (Metabolism and nutrition disorders) | 24 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 0
Dizziness (Nervous system disorders) | 23 | 0
Dysgeusia (Nervous system disorders) | 7 | 0
Headache (Nervous system disorders) | 21 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Syncope (Nervous system disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 4 | 0
Confusional state (Psychiatric disorders) | 5 | 0
Depression (Psychiatric disorders) | 15 | 0
Insomnia (Psychiatric disorders) | 12 | 0
Chromaturia (Renal and urinary disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 5 | 0
Haematuria (Renal and urinary disorders) | 7 | 0
Nephrolithiasis (Renal and urinary disorders) | 7 | 0
Pollakiuria (Renal and urinary disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 0
Rash (Skin and subcutaneous tissue disorders) | 32 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 7 | 0
Hypertension (Vascular disorders) | 9 | 0
Hypotension (Vascular disorders) | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes